CLINICAL TRIAL: NCT05383534
Title: To Study the Pharmacokinetic and Cardiovascular Effects of Propofol With Respect to Pharmacogenetics in the Pakistani Population.
Brief Title: To Study the Pharmacokinetic and Cardiovascular Effects of Propofol With Respect to Pharmacogenetics in Pakistani Population
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Collaborators: Holy Family Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Uzma Naeem, Associate Professor, Riphah International University
Other Study IDs: Riphah/IIMC/IRC/20/002
Record Dates: First submitted 2022-05-16; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Healthy Volunteer
Keywords: Pakistani population, Propofol serum concentration, adverse effects.
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Propofol Injection — propofol injections were used for the induction of anesthesia according to the body weight of the patients.

SUMMARY:
This study aimed to determine the effects of genetic variabilities among the Pakistani population on propofol serum concentration and its adverse effects mainly cardiovascular adverse effects. cardiovascular adverse effects are the main concern for the anesthetists, if a person is genetically more prone to these adverse effects it can be lethal for that.

DETAILED DESCRIPTION:
Propofol is a phenolic byproduct, available as an oil-in-water intravenous emulsion for calming and mesmerizing purposes. It is among the most widely used intravenous soporific drugs that are used for induction and maintenance of general anesthesia, procedural calmness, and to gain tranquility in ICU patients. Advantages of propofol include easy control of the depth of anesthesia, rapid recovery of consciousness, and less postoperative nausea and vomiting. Due to these characteristics, propofol has turned out to be the standard agent for induction of anesthesia. Although it is safe, it doesn't mean that it is devoid of any adverse effects. Important adverse effects of propofol include cardiovascular effects, mild respiratory depression, bronchospasm in patients with reactive airways, pain on the injection site, and rarely myoclonus. The most common cardiovascular effects are hypotension and bradycardia. These cardiovascular effects are produced by propofol-induced suppression of sympathetic activity, inhibitory effects on the baroreceptor reflex, stimulation of nitric oxide-mediated vasodilation, and blockage of voltage-gated sodium and potassium channel.

However, in clinical practice, a large inter-individual variability is observed in response to this anesthetic. Concerning the effectiveness, standard dose, and harmful drug responses of propofol, genetic variations have been appraised to add about 20%-30% to this variability and it is due to variations in allele frequencies. These genotype frequencies have been studied in many racial populations and they were found to be correlated with variation in drug responses. Most of these studies have been practiced determining the pharmacogenetic information for better pharmaceutical care, by preventing therapeutic collapse or critical adverse reactions in a population linked to this genetic variability. These inter-individual differences in genotype frequencies affect the efficiency of enzymes that are required for the metabolism of propofol. This change in the metabolic rate of this drug necessitates the modifications in the optimum dose required for effective general anesthesia with minimum adverse effects.

Propofol is primarily metabolized in the liver by cytochrome P450 2B6 (CYP2B6), cytochrome P450 2C9 (CYP2C9), and by UDP-glucuronosyltransferase 1A9 (UGT1A9). It is suggested that single nucleotide polymorphisms in the genes coding for these enzymes can be accountable for the inter-individual variations of propofol response. This can lead to unpredictable effects even with the recommended doses of propofol. The most common functionally deficient allele is CYP2B6*6 (c.516) G>T rs3745274 and (c.785) A>G rs2279343), which occurs at frequencies of 15 to over 60% in different populations. These alleles are accountable for the low CYP2B6 expression phenotype and are found to be associated with enhanced plasma levels of propofol. For the CYP2C9 gene, more than sixty-five haplotypes have been described, but in global studies, only two non-synonymous changes, (c.430C>T, rs1799853, CYP2C9*2) and (c.1075A>C, rs1057910, CYP2C9*3) are intensively analyzed. These two are found to be associated with low enzymatic activity and so raised serum levels of propofol.

Concerning the Pakistani population, the prevalence of variant allele c.785A>G, rs2279343 is 48% and 36% of c.516G>T, rs3745274 allele. These two alleles are linked with decreased activity of the CYP2B6 enzyme. The frequent alleles of CYP2C9 in Pakistani population are c.1075A>C, rs1057910 and rs1799853, c.430C > T, their frequencies are 10% & 7% respectively. Genetic testing suggested that around 30% Pakistani population has some level of compromised CYP2C9 function. So, the individuals with these genetic polymorphisms need modification in the induction and maintenance dose of the propofol because in normal doses the slow metabolism of propofol can lead to more intense cardiovascular effects and other adverse effects produced by the propofol. The effect of these variant alleles on propofol pharmacokinetics and adverse effect profile is not studied to date in the Pakistani population, so this study will verify this. Awareness of the consequences of important changes in the CYP2B6 and CYP2C9 genes in propofol metabolism would make it possible to increase the safety of patients undergoing general intravenous anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Pakistani individuals between ages 18-60 years undergoing elective surgeries (Open/Laparoscopic guided) induced with propofol.
* Patients in classes I and II of the American Society of Anesthesiologists (ASA) scale.

Exclusion Criteria:

* Not of Pakistani origin

  * Extremes of age
  * Patients in classes III, IV, V &, VI of the ASA scale.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: study population contained patients of Pakistani origin.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
genetic variabilities in propofol metabolism among the Pakistani population and its relationship with serum propofol levels, and propofol related adverse effects | one year
  genetic variabilities among the Pakistani population at the enzymatic level can affect the propofol metabolism and so the adverse effects profile especially the cardiovascular adverse effects. these cardiovascular effects are expressed in the form of mean blood pressure and heart rate. if the dose of propofol is calculated according to the genetic makeup of the individual chances of severe drug-related cardiovascular adverse effects can be decreased.

CONTACTS AND LOCATIONS:
Locations (1):
- Uzma Naeem, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naeem U, Waheed A, Azeem Y, Awan MN. Effects of body mass index on propofol-induced cardiovascular depression in the Pakistani population. Pak J Med Sci. 2023 Mar-Apr;39(2):534-538. doi: 10.12669/pjms.39.2.6787. PMID 36950415